CLINICAL TRIAL: NCT06028217
Title: A Prospective Study on Pathogen Investigation, Risk Factors, and Prognostic Factors Analysis of Hospital Acquired Pneumonia (HAP)
Brief Title: Chinese Hospital Acquired Pneumonia Collaboration Network: Epidemiology, Diagnosis and Treatment
Acronym: CHAPTER
Status: Not yet recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Jieming QU, Professor, Ruijin Hospital
Other Study IDs: CHAPTER-1.7
Record Dates: First submitted 2023-08-31; First posted 2023-09-08 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-08

CONDITIONS: Hospital-acquired Pneumonia; Antibiotic Resistant Infection
MeSH Terms: conditions — Healthcare-Associated Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- survival group: patients still survive at 28 days
  Interventions: Other: prognosis status
- mortality group: patients die within 28 days
  Interventions: Other: prognosis status

INTERVENTIONS:
Other: prognosis status — observatory; patients will be divided into survival group and mortality group according to their prognosis at day 28

SUMMARY:
The goal of this prospective and observatory study is to learn about the pathogen, clinical manifestations, prognosis, treatment and antibiotic resistance of bacteria in hospital-acquired pneumonia patients in China.

The main purposes of this study are:

1. clarify the regional differences and changes over time in the pathogen spectrum and antibiotic resistance rate among HAP patients in China;
2. build a continuously optimized nationwide HAP pathogen and antibiotic resistance surveillance network;
3. identify the molecular epidemiology of common pathogens

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old.
2. Meets the clinical diagnostic criteria for HAP in the 2018 HAP/VAP guidelines. Chest X-ray or CT shows new or progressive infiltrative shadows, consolidation shadows, or ground glass shadows, combined with 2 or more of the following 3 clinical symptoms, to establish a clinical diagnosis: 1) Fever, body temperature>38 ℃; 2) Purulent airway secretions; 3) Peripheral blood white blood cell count >10 × 10^9/L or <4 × 10^9/L.
3. Having qualified evidence of responsible pathogen. On the basis of clinical diagnosis, one of the following conditions should be met simultaneously: 1) Qualified lower respiratory tract secretions (neutrophil count >25/low magnification field, epithelial cell count <10/low magnification field, or a ratio of the two >2.5:1), pathogenic bacteria cultured through bronchoscopy anti pollution brush (PSB), bronchoalveolar lavage fluid (BALF), lung tissue or sterile body fluid, and consistent with clinical manifestations; 2) Pathology, cytopathology, or direct microscopic examination of lung tissue specimens showing fungi and evidence of tissue damage; 3) The serum IgM antibodies of atypical pathogens or viruses change from negative to positive, or the titers of specific IgG antibodies in both acute and recovery phases show a 4-fold or more change. During the outbreak of respiratory viruses and with a history of epidemiological contact, respiratory secretions were tested positive for corresponding virus antigens, nucleic acid tests, or virus culture.
4. obtained informed consent

Exclusion Criteria:

1. Those who cannot understand and execute the investigation plan.
2. Active pulmonary tuberculosis;
3. Severely immunosuppressed patients: absolute neutrophil count <0.5× 10^9/L, CD4<200/ml.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hospital-acquired pneumonia adult patients with qualified evidence of responsible pathogen in China
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
mortality at day 28 | 28 days after enrollment
  prognosis

SECONDARY OUTCOMES:
clinical characteristics | 0 day, 3 days, 7days, 14 days and 28 days after enrollment
  symptoms, physical examinations, comorbidity, laboratory tests, imaging findings and treatment
pathogen | 0 day, 3 days, 7days, 14 days and 28 days after enrollment
  molecular characteristics of responsible pathogen; antibiotic resistance of bacteria